CLINICAL TRIAL: NCT02199496
Title: An Open-Label Phase I/II Pilot Study to Assess the Safety/Tolerability and Efficacy of Ustekinumab for Symptomatic Gastrointestinal Inflammation Associated With Common Variable Immunodeficiency
Brief Title: Study of Safety, Tolerability, and Efficacy of Ustekinumab for Symptomatic Gastrointestinal Inflammation Associated With Common Variable Immunodeficiency
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140153; 14-I-0153
Record Dates: First submitted 2014-07-23; First posted 2014-07-24 (Estimated); Results first posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-07

CONDITIONS: Gastrointestinal Inflammation Associated With CVID; CVID Enteropathy
Keywords: Malabsorption; Enteropathy; Diarrhea; IL-12
MeSH Terms: conditions — Malabsorption Syndromes; Intestinal Diseases; Diarrhea | interventions — Ustekinumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Ustekinumab-Single-dose Phase 1, Multi-dose Phase 2 (Experimental): Subjects given an induction dose of 270 mg Stelara (ustekinumab) subcutaneously then re-enrolled into the multi-dose phase. In multi-dose phase, subjects given an induction dose of 270 mg Stelara (ustekinumab) subcutaneously followed by every 8 week maintenance doses of 90 mg Stelara (ustekinumab) subcutaneously at week 8, week 16, week 24, week 32, and week 40
  Interventions: Biological: Stelara (ustekinumab)
- Cohort 2: Ustekinumab-Multi-dose Phase 2 (Experimental): Subjects given an induction dose of 270 mg Stelara (ustekinumab) subcutaneously followed by every 8 week maintenance doses of 90 mg Stelara (ustekinumab) subcutaneously at week 8, week 16, week 24, week 32, and week 40
  Interventions: Biological: Stelara (ustekinumab)

INTERVENTIONS:
Biological: Stelara (ustekinumab) — * In the single-phase part of the study, subjects receive a single dose of Stelara (ustekinumab) 270 mg subcutaneously on Day 0 study visit.
  * In the multi-phase part of the study, subjects receive single dose of Stelara (ustekinumab) 270 mg subcutaneously on Day 0 study visit with follow up dose of Stelara (ustekinumab) 90 mg subcutaneously at Week 8, Week 16, Week 24, Week 32 and Week 40

SUMMARY:
Background:

- Some people with Common Variable Immunodeficiency Disease (CVID) have gastrointestinal inflammation. This can cause diarrhea, weight loss, and not being able to absorb nutrition from food. Researchers want to see if the drug ustekinumab can help these problems. This drug blocks some proteins that cause inflammation.

Objective:

- To test the safety and efficacy of the drug ustekinumab for people with CVID with gastrointestinal inflammation.

Eligibility:

- Adults ages 18-75 with CVID. They must have chronic diarrhea, have unintentionally lost weight in the last year, and/or need to use nutritional supplements to maintain their weight.

Design:

Participants will undergo the following screening studies to make sure that this study is a good fit for your medical situation, and to make sure it is safe for you to receive the study medications tests, including tests for HIV and hepatitis . This will be done as an inpatient at the NIH Clinical Center and takes about 5-6 days:

* Participants will be screened with:
* Medical history
* Physical exam
* Blood tests, including tests for HIV and hepatitis.
* Stool tests, including a timed 48 hour collection for fat malabsorption and a 24 hour collection for protein malabsorption
* Urine tests, including a pregnancy test for any women with the ability to have a child
* Chest CT scan to look for infection
* D-xylose testing, which involves drinking a sugary solution and then having a blood sample drawn to test carbohydrate (sugar) malabsorption
* Hydrogen breath testing for test for small intestinal bacterial overgrowth (SIBO) this test also involves drinking a sugary solution and then collecting breath samples
* Upper endoscopy (EGD) and/or colonoscopy to look at the lining of the GI tract and take biopsies for testing. This will be done under sedation by a qualified gastroenterologist.

Participants who complete screening and meet all criteria will then return to the NIH Clinical Center for the following visits:

* First Treatment Visit (1 clinic day): Medical history, physical exam, measurement of vital signs and weight, review of medications, and an assessment of number and consistency of stools each day. A pregnancy test for women of childbearing potential. A nurse will give you three shots of 90 mg ustekinumab (270 mg total dose) by very small needles injected under the skin, and then observe you for 1 hour.
* Week 8 Treatment Visit (1 clinic day): Medical history, physical exam, measurement of vital signs and weight, review of medications, and an assessment of number and consistency of stools each day. Blood, urine and stool samples will be collected. A pregnancy test for women of childbearing potential. A nurse will give you one 90 mg dose of ustekinumab by a very small needle injected under the skin, and then observe you for 1 hour.
* Week 16 Treatment Visit (1 clinic day): Medical history, physical exam, measurement of vital signs and weight, review of medications, and an assessment of number and consistency of stools each day. Blood, urine and stool samples will be collected. A pregnancy test for women of childbearing potential. A nurse will give you one 90 mg dose of ustekinumab by a very small needle injected under the skin, and then observe you for 1 hour.
* Week 24 Treatment and Mid-point Evaluation Visit (4-6 inpatient days): Medical history, physical exam, measurement of vital signs and weight, review of medications, and an assessment of number and consistency of stools each day. Blood, urine and stool samples will be collected, including repeating the d-xylose carbohydrate malabsorption testing, the 24 hour stool collection for protein malabsorption and the 48 hour stool collection for fat malabsorption. A pregnancy test for women of childbearing potential. A nurse will give you one 90 mg dose of ustekinumab by a very small needle injected under the skin, and then observe you for 1 hour.
* Week 32 Treatment Visit: Medical history, physical exam, measurement of vital signs and weight, review of medications, and an assessment of number and consistency of stools each day. Blood, urine and stool samples will be collected. A pregnancy test for women of childbearing potential. A nurse will give you one 90 mg dose of ustekinumab by a very small needle injected under the skin, and then observe you for 1 hour.
* Week 40 Treatment Visit: Medical history, physical exam, measurement of vital signs and weight, review of medications, and an assessment of number and consistency of stools each day. Blood, urine and stool samples will be collected. A pregnancy test for women of childbearing potential. A nurse will give you one 90 mg dose of ustekinumab by a very small needle injected under the skin, and then observe you for 1 hour.
* Week 48 ...

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety/tolerability and efficacy of using ustekinumab in subjects with common variable immunodeficiency CVID or selective IgG subclass deficiency (functional agammaglobulinemia) who have associated symptomatic gastrointestinal inflammation (CVID enteropathy). Ustekinumab (a Food and Drug Administration [FDA] approved drug) is a monoclonal antibody to interleukin (IL)-12/23p40. CVID is a clinically heterogeneous disorder characterized by decreased serum immunoglobulin IgG and IgA levels. In addition to chronic or recurrent pyogenic sino-pulmonary infections, many patients develop non-infectious gastrointestinal manifestations that can be disabling or fatal. Currently there is no standard therapy for the associated gastrointestinal disease outside of empiric nutritional intervention for weight loss, anti-diarrheal agents, and non-specific anti-inflammatory agents.

Recently, gut inflammation complicating functional hypogammaglobulinemia due to CVID and selective IgG subclass deficiency has been characterized as a T helper type 1 (Th1) inflammatory response, with excess IL-12 cytokine production associated with diarrhea and weight loss as well as reduced D-xylose absorption and steatorrhea. This protocol aims to test specific anti-IL-12 therapy in this patient group. It has been previously shown that therapy targeted to IL-12 successfully treated the Th1 gut inflammation of Crohn s disease (CD). Ustekinumab, a monoclonal antibody to the p40 subunit of IL-12 and IL-23, is FDA approved for the treatment of moderate to severe plaque psoriasis, active psoriatic arthritis, and more recently, moderately to severely active CD. This protocol is designed to measure the safety of ustekinumab in patients with functional hypogammaglobulinemia and CVID enteropathy, as well as measure effects on symptoms, gut function, expression of immune cell surface markers, production of cytokines and global gene expression from blood and gut mucosal mononuclear cells, and the gut microbiota.

Patients with CVID and selective IgG subclass deficiency with gastrointestinal symptoms of malabsorption, maldigestion, and chronic diarrhea will be enrolled into this study. Subjects (up to a total of 10 individuals) will receive a treatment dose of 270 mg (3 doses of 90 mg either single-use prefilled syringe or single-use vial, depending on availability) will be injected subcutaneously in subjects by qualified nursing staff on the Day 0 study visit. Subjects will then receive a follow up treatment dose of 90 mg at Week 8, Week 16, Week 24, Week 32 and Week 40 and be followed for a total of 48 weeks.

Subjects will have study procedures prior to treatment and 48 weeks post-treatment, these include upper and/or lower endoscopies, to measure changes in immune responses and studies to evaluate physiologic measures of gut function at 48 weeks, as well as routine safety monitoring throughout the study. Gut absorption tests will be performed at the Week 24 visit. Variables will include safety (adverse event rate), clinical (weight, stool frequency, results of gut absorption tests), and laboratory (lymphocyte and cytokine assays) parameters for descriptive summary statistical analysis (n, mean, median, standard deviation, minimum and maximum range).

ELIGIBILITY:
* DIAGNOSIS AND CRITERIA FOR INCLUSION:

A subject is eligible for the study if all of the following criteria are met:

* Has given written informed consent.
* Is male or female aged 18 through 75 years.
* Has CVID or selective IgG subclass deficiency of either one or concomitant IgG subclasses comprising IgG1, IgG2, IgG3 or IgG4 (functional hypogammaglobulinemia) diagnosed prior to screening as based on the International Union of Immunological Societies (IUIS) criteria.
* Has a documented, unintended loss of >5% of their body weight over the last year or requires nutritional supplements to maintain his/her body weight and/or has chronic diarrhea defined as a complaint of at >/= 50% of stools are non-formed for at least 4 consecutive weeks per patient history. Alternately, must be dependent on a therapeutic dose of antidiarrheals (e.g., loperamide or diphenoxylate with atropine) for control of chronic diarrhea.
* If taking oral antibiotics chronically, must have used a stable dose of the antibiotic continuously for at least 2 weeks prior to start of screening period.
* Is willing to have samples stored.
* Be willing to consistently take appropriate measures to avoid pregnancy through the Week 48 study point. All subjects will be informed of the potential risks of ustekinumab during pregnancy and counseled on pregnancy avoidance appropriate to the subject s circumstances (e.g. fertility status, medical contraindications to hormonal birth control, and/or personal or religious beliefs regarding pregnancy avoidance). Subject to the judgment and discretion of the PI, some subjects may not need to take pregnancy

avoidance measures. Patient handout on pregnancy avoidance will be provided to patients at the time of consent and discussion regarding pregnancy avoidance during the study.

-Subjects who have previously been treated with a single 270 mg dose of ustekinumab on this study must be greater than 6 months from their treatment dose and have had recurrence of enteropathy symptoms.

CRITERIA FOR EXCLUSION:

A subject is excluded from the study if any of the following criteria are met:

GENERAL CRITERIA:

* Has any clinically significant disease or condition (e.g., renal, hepatic, neurological, cardiovascular, pulmonary, endocrinologic, psychiatric, hematologic, urologic, or other acute or chronic illness) that in the opinion of the investigator would make the subject an unsuitable candidate for this trial, or put the subject at undue risk by participating in this study.
* Is a woman who has a positive pregnancy test or who is breast-feeding
* Is a woman who does not agree to abide by the contraceptive measures required to prevent pregnancy during participation in the study, or meets exemption criteria for contraceptive measures, as outlined in the protocol.
* Has any of the following clinical chemistry values:

  * AST >2.5 times upper limit of normal (ULN).
  * ALT >2.5 times ULN.
  * Serum bilirubin >1.5 times ULN.
  * Serum creatinine >1.5 times ULN.
  * Alkaline phosphatase >2.5 times ULN.
* Has a hemoglobin level <9 g/dL or hematocrit <30%.
* Has an International Normalized Ratio (INR) >1.3 or a Partial Thromboplastin Time (PTT) >3 sec of ULN.
* Has the following cell counts (cells/microL):

  * Platelet count <75,000 or >800,000.
  * White blood cell count <2,000.
  * Neutrophil count <1,000.
* Has a current infection requiring intravenous antibiotics, a serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., pneumonia, septicemia).
* Has a history of cancer within the past 5 years, with the exception of excised basal cell carcinoma, squamous cell carcinoma of the skin, or cervical carcinoma in situ.
* Had a dependency for any illicit drug, chemical, or alcohol within the past 5 years.
* Has a history of active tuberculosis (TB) (or a chest x-ray (CXR) with findings suggestive of old TB infection including calcified nodular lesions, apical fibrosis, or pleural scarring), acute or chronic hepatitis B, hepatitis C, human immunodeficiency virus (HIV) or opportunistic infections.

GASTROINTESTINAL CRITERIA

-Has a stool sample determined positive for acute gastrointestinal infection with impact of occurrence on gastrointestinal inflammation as determined by principal investigator during screening. In addition, stool samples positive for GI pathogens will be discussed with an infectious disease physician to determine impact of occurrence on gastrointestinal inflammation. If organism thought to be pathogenic, the subject will be treated with appropriate therapy. This will be documented in the subject s medical record.

PRIOR MEDICATION CRITERIA

* Received daily corticosteroids within 1 month prior to receiving study agent. The use of short-term or single-dose corticosteroids as a pretreatment regimen for IVIG is acceptable.
* Received any investigational drug within 3 months prior to receiving study agent.
* Received certolizumab or natalizumab within 3 months prior to receiving study agent
* Received vedolizumab, infliximab, etanercept, or adalimumab within 2 months prior to receiving study agent.
* Received cyclosporine, tacrolimus, sirolimus, pimecrolimus, mycophenolate mofetil or any other systemic immunosuppressants within 1 month prior to receiving study agent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2020-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan J Fuss, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Cunningham-Rundles C, Bodian C. Common variable immunodeficiency: clinical and immunological features of 248 patients. Clin Immunol. 1999 Jul;92(1):34-48. doi: 10.1006/clim.1999.4725. PMID 10413651
- [Background] Sandborn WJ, Gasink C, Gao LL, Blank MA, Johanns J, Guzzo C, Sands BE, Hanauer SB, Targan S, Rutgeerts P, Ghosh S, de Villiers WJ, Panaccione R, Greenberg G, Schreiber S, Lichtiger S, Feagan BG; CERTIFI Study Group. Ustekinumab induction and maintenance therapy in refractory Crohn's disease. N Engl J Med. 2012 Oct 18;367(16):1519-28. doi: 10.1056/NEJMoa1203572. PMID 23075178
- [Background] Mannon PJ, Fuss IJ, Dill S, Friend J, Groden C, Hornung R, Yang Z, Yi C, Quezado M, Brown M, Strober W. Excess IL-12 but not IL-23 accompanies the inflammatory bowel disease associated with common variable immunodeficiency. Gastroenterology. 2006 Sep;131(3):748-56. doi: 10.1053/j.gastro.2006.06.022. PMID 16952544
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-I-0153.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Single-dose Phase 1, Multi-dose Phase 2: Subjects given single dose of 270mg Ustekinumab subcutaneously then re-enrolled into the multi-dose phase. In multi-dose phase subjects given single dose of 270mg Ustekinumab subcutaneously with follow up treatment doses of 90 mg (1 dose of 90 mg) at week 8, week 16, week 24, week 32, and week 40
- Cohort 2: Multi-Dose Ustekinumab Phase 2: Subjects given single dose of 270mg Ustekinumab subcutaneously then follow up treatment doses of 90 mg (1 dose of 90 mg) at week 8, week 16, week 24, week 32, and week 40
Period: Ustekinumab-Single Dose
Arm/Group | Cohort 1: Single-dose Phase 1, Multi-dose Phase 2 | Cohort 2: Multi-Dose Ustekinumab Phase 2
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0
Period: Ustekinumab-Multi-dose
Arm/Group | Cohort 1: Single-dose Phase 1, Multi-dose Phase 2 | Cohort 2: Multi-Dose Ustekinumab Phase 2
Started | 3 | 2 (Cohort 2 only participated in multi-dose phase 2)
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Ustekinumab-Single-dose Phase 1, Multi-dose Phase 2 | Cohort 2: Ustekinumab-Multi-dose Phase 2 | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Increase in Infection or Serious Adverse Events (SAEs) Related to Single Dose Administration of Ustekinumab
Description: Whether treatment with ustekinumab is safe and tolerated in patients with common variable immunodeficiency (CVID) enteropathy as determined by no significant increase in infection or serious adverse events
Time Frame: 6 months
Population: Participants who received ustekinumab
Measure: Number; unit: participants
Groups:
- Cohort 1: Ustekinumab-Single Dose Phase 1: Single dose of 270mg ustekinumab subcutaneously
Arm/Group | Cohort 1: Ustekinumab-Single Dose Phase 1
Number analyzed (Participants) | 3
participants | 0

2. Primary Outcome: Number of Participants With Increase in Infection or Serious Adverse Events (SAEs) Related to Multi-dose Administration of Ustekinumab (Cohort 1)
Description: as for outcome 1
Time Frame: 48 weeks
Population: Participants who received ustekinumab
Measure: Number; unit: participants
Groups:
- Cohort 1: Ustekinumab-Multi-dose Phase 2: Single dose of 270mg ustekinumab subcutaneously then follow up doses of 90 mg ustekinumab subcutaneously at week 8, week 16, week 24, week 32, and week 40
Arm/Group | Cohort 1: Ustekinumab-Multi-dose Phase 2
Number analyzed (Participants) | 3
participants | 0

3. Primary Outcome: Number of Participants With Increase in Infection or Serious Adverse Events (SAEs) Related to Multi-dose Administration of Ustekinumab (Cohort 2)
Description: as for outcome 1
Time Frame: 48 weeks
Population: Participants who received ustekinumab
Measure: Number; unit: participants
Groups:
- Cohort 2: Ustekinumab-Multi-dose Phase 2: Single dose of 270mg ustekinumab subcutaneously then follow up doses of 90 mg ustekinumab subcutaneously at week 8, week 16, week 24, week 32, and week 40
Arm/Group | Cohort 2: Ustekinumab-Multi-dose Phase 2
Number analyzed (Participants) | 2
participants | 0

ADVERSE EVENTS:
Time Frame: 6 months for Phase 1 and 48 Weeks for Phase 2
Arm/Group | Cohort 1: Ustekinumab-Single Dose Phase 1 | Cohort 1: Ustekinumab-Multi-dose Phase 2 | Cohort 2: Ustekinumab-Multi-dose Phase 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 2/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Ustekinumab-Single Dose Phase 1 (N=3) | Cohort 1: Ustekinumab-Multi-dose Phase 2 (N=3) | Cohort 2: Ustekinumab-Multi-dose Phase 2 (N=2)
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Ustekinumab-Single Dose Phase 1 (N=3) | Cohort 1: Ustekinumab-Multi-dose Phase 2 (N=3) | Cohort 2: Ustekinumab-Multi-dose Phase 2 (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 0 | 1
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 0 | 1
Rectal tenesmus (Gastrointestinal disorders) | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1
Chills (General disorders) | 1 | 1 | 0
Fatigue (General disorders) | 1 | 2 | 0
Injection site pain (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 1
Oedema (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Swelling (General disorders) | 0 | 0 | 1
Tenderness (General disorders) | 0 | 0 | 2
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 1 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0
Enterovirus infection (Infections and infestations) | 1 | 1 | 0
Gastroenteritis Escherichia coli (Infections and infestations) | 0 | 3 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 1 | 0
Gastrointestinal bacterial overgrowth (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 1
Alpha-1 anti-trypsin increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Blood 1,25-dihydroxycholecalciferol increased (Investigations) | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 1
Blood chloride increased (Investigations) | 1 | 1 | 0
Blood copper decreased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
Blood glucose decreased (Investigations) | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 2
Blood iron decreased (Investigations) | 0 | 1 | 1
Blood lactate dehydrogenase (Investigations) | 2 | 1 | 1
Blood urea increased (Investigations) | 0 | 0 | 1
Blood zinc decreased (Investigations) | 0 | 1 | 1
Body temperature increased (Investigations) | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0
Clostridium test positive (Investigations) | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 2 | 1
Epstein-Barr virus test positive (Investigations) | 0 | 0 | 1
Faecal calprotectin increased (Investigations) | 0 | 1 | 0
Faecal fat increased (Investigations) | 0 | 1 | 0
False positive investigation result (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0
Haematocrit decreased (Investigations) | 1 | 2 | 1
International normalised ratio increased (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 2 | 0
Norovirus test positive (Investigations) | 1 | 2 | 0
Platelet count decreased (Investigations) | 1 | 1 | 1
Prothrombin time prolonged (Investigations) | 2 | 0 | 0
Prothrombin time shortened (Investigations) | 0 | 1 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 1
Vitamin B6 increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 2 | 3 | 0
White blood cells urine positive (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 3 | 0
Vitamin B6 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Vitamin E deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Nightmare (Psychiatric disorders) | 0 | 1 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT02199496/Prot_SAP_000.pdf